CLINICAL TRIAL: NCT04963426
Title: Empowering Adolescents to Lead Change Using Health Data
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: World Health Organization (Other)
Collaborators: Fondation Botnar (Unknown); University of Bern (Other); University of Wollongong (Other)
Responsible Party: Principal Investigator, Regina Guthold, Scientist, World Health Organization
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ERC.0003397
Record Dates: First submitted 2021-07-05; First posted 2021-07-15 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: adolescent health; students; schools; risk factors; protective factors; school health services
MeSH Terms: interventions — Protective Factors; Drug Delivery Systems

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): The intervention consists of interactive workshops that will be facilitated by WHO and trained local personnel and involve students, teachers and local authorities. In the workshops, the Global Accelerated Action for the Health of Adolescents (Global AA-HA!) approach will be used to:
  * identify adolescent health needs through exploring the collected baseline data;
  * assess policies and practices already in place;
  * identify gaps and needs for action to improve health. A menu of actions will be identified, prioritized, implemented and monitored.
  Interventions: Behavioral: Behavioral interventions targeting multiple risk behaviors as well as protective factors; Other: School-level interventions targeting the school environment and system
- Control arm (No Intervention): The schools in the control arm will not participate in any intervention and continue 'as usual' after the baseline surveys.

INTERVENTIONS:
Behavioral: Behavioral interventions targeting multiple risk behaviors as well as protective factors — Depending on the baseline data and prioritization of actions, behavioral interventions related to the following topics will be implemented: alcohol use, dietary behaviors, drug use, hygiene, mental health, physical activity, protective factors, sexual behaviors, tobacco use, violence and unintentional injury.
  Arms: Intervention arm
Other: School-level interventions targeting the school environment and system — Depending on the baseline data and prioritization of actions, and based on the Global Standards for Health Promoting Schools, school-level interventions related to the following will be implemented: school policies and resources, school governance and leadership, school and community partnerships, school curriculum, school social-emotional environment, school physical environment, school health services
  Arms: Intervention arm

SUMMARY:
This study is a cluster randomized trial carried out in schools of secondary cities of four low- and middle income countries. Baseline surveys in 30 randomly selected schools will assess the health behaviours of 13-17 year old students as well as school policies and practices. The intervention arm (15 schools) will use the baseline information to develop a package of actions in collaboration with students, teachers, and local authorities that will subsequently be implemented an monitored over two years. Follow-up surveys to evaluate the effectiveness of the implemented actions will be conducted after two years in all 30 previously selected schools.

DETAILED DESCRIPTION:
The objective of this study is to generate health information through school surveys and use this information directly and locally, involving adolescents, to change policies and plan programmes to improve health.

The study is carried out in secondary cities of four low- and middle income countries, including Sekondi-Takoradi, Ghana; Jaipur, India; Spanish Town, Jamaica; and Fez, Morocco.

In each of the four cities, 30 schools are randomly selected. Baseline surveys will be conducted to assess (1) 13-17 year old student's health behaviours using the Global School-based Student Health Survey (GSHS); and (2) health policies and practices in the selected schools using the Global School Health Policies and Practices Study (G-SHPPS). Additionally, the physical activity module of the GSHS questionnaire will be validated against objective measurement devices in one randomly selected class of 15 randomly selected schools.

Schools will be randomly allocated to the intervention (15 schools) or control arm (15 schools) of the study. The intervention group will participate in interactive workshops using the Global Accelerated Action for the Health of Adolescents (Global AA-HA!) approach and the framework of Making every school a health-promoting school to:

1. Identify adolescent health needs through exploring the collected data;
2. Assess policies and practices already in place;
3. Identify gaps and needs for action to improve health. Students, teachers and local authorities will propose and prioritize policy and programme solutions from menus of effective interventions for school-, community- or city-level implementation, supported by the Ministries of Health and Education and WHO.

Repeat GSHS and G-SHPPS surveys will be conducted two years later in all schools to assess effectiveness of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* School going
* Aged 13-17 years

Exclusion Criteria:

* Not going to school
* Outside the age range 13-17 years

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12612 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Alcohol use | Two years
  Self-reported alcohol use measured with the Global School-based Student Health Survey (GSHS)
Dietary behaviors | Two years
  Self-reported dietary behaviors measured with the Global School-based Student Health Survey (GSHS)
Drug use | Two years
  Self-reported drug use measured with the Global School-based Student Health Survey (GSHS)
Hygiene | Two years
  Self-reported hygiene measured with the Global School-based Student Health Survey (GSHS)
Mental health | Two years
  Self-reported mental health measured with the Global School-based Student Health Survey (GSHS)
Physical activity | Two years
  Self-reported physical activity measured with the Global School-based Student Health Survey (GSHS)
Protective factors | Two years
  Self-reported protective factors measured with the Global School-based Student Health Survey (GSHS)
Sexual behaviors | Two years
  Self-reported sexual behaviors measured with the Global School-based Student Health Survey (GSHS)
Tobacco use | Two years
  Self-reported tobacco use measured with the Global School-based Student Health Survey (GSHS)
Violence and unintentional injury | Two years
  Self-reported violence and unintentional injury measured with the Global School-based Student Health Survey (GSHS)

OTHER OUTCOMES:
School-level policies and practices | Two years
  School-level outcomes related to the following: school policies and resources, school governance and leadership, school and community partnerships, school curriculum, school social-emotional environment, school physical environment, school health services measured with the Global School Health Policies and Practices Study (G-SHPPS)

CONTACTS AND LOCATIONS:
Overall Officials: Regina Guthold, PhD, Principal Investigator — World Health Organization
Locations (5):
- WHO, Sekondi-Takoradi, Ghana
- WHO, Jaipur, India
- WHO, Spanish Town, Jamaica
- WHO, Fes, Morocco
- WHO, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
After a two year window following completion of data collection, the GSHS and G-SHPPS data will be released as public access datasets, including in the WHO NCD microdata repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The documents above will become available after the study protocol has been published in a scientific journal.

REFERENCES:
- [Derived] Guthold R, Kann L, Bhatti L, Abduvahobov P, Ansong J, Atkinson U, Baltag V, Caffe S, Caixeta R, Diallo CB, Fouad H, Haddad S, Hachri H, Jaggi JA, Joshi P, Karna P, Louazani SA, Mbola Mbassi S, Mehta R, Mudgal Y, Nigg CR, Okely AD, Ondarsuhu D, Ouaourir T, Trhari FZ, Riley LM. Effectiveness of a participatory approach to develop school health interventions in four low resource cities: study protocol of the 'empowering adolescents to lead change using health data' cluster randomised controlled trial. BMJ Open. 2023 Jul 5;13(7):e071353. doi: 10.1136/bmjopen-2022-071353. PMID 37407059